CLINICAL TRIAL: NCT01350271
Title: Comparative Efficacy of Different Mebendazole Polymorphs in the Treatment of Soil-transmitted Helminth Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kelaniya (Other)
Responsible Party: Principal Investigator, N R de Silva, Professor of Parasitology, University of Kelaniya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P39/04/2010; Ragama ERC (Registry Identifier: www.clinicaltrials.org)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Necator Americanus Infection
Keywords: Hookworm; Necator americanus; Mebendazole
MeSH Terms: conditions — Ancylostomiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo tablets produced by the State Pharmaceutical Manufacturing Corporation of Sri Lanka
  Interventions: Drug: Placebo
- Mebendazole polymorph A and C 500 mg (Active Comparator): Mebendazole tablets produced by the State Pharmaceutical Manufacturing Corporation of Sri Lanka, containing 500mg of mebendazole as a 50:50 mixture of Polymorphs A and C
  Interventions: Drug: Mebendazole polymorph A and C 500 mg
- Mebendazole polymorph C 500 mg (Experimental): Mebendazole tablets manufactured by the State Pharmaceutical Manufacturing Corporation of Sri Lanka, containing 500mg dose of mebendazole as Polymorph C alone
  Interventions: Drug: Mebendazole polymorph C

INTERVENTIONS:
Drug: Mebendazole polymorph A and C 500 mg — Mebendazole tablets produced by the State Pharmaceutical Manufacturing Corporation of Sri Lanka, containing 500mg of mebendazole as a 50:50 mixture of Polymorphs A and C
  Other Names: Lot FG10M01
  Arms: Mebendazole polymorph A and C 500 mg
Drug: Mebendazole polymorph C — Mebendazole tablets manufactured by the State Pharmaceutical Manufacturing Corporation of Sri Lanka, containing 500mg dose of mebendazole as Polymorph C alone
  Other Names: Lot FG10H01
  Arms: Mebendazole polymorph C 500 mg
Drug: Placebo — Placebo tablets produced by the State Pharmaceutical Manufacturing Corporation of Sri Lanka
  Arms: Placebo

SUMMARY:
Mebendazole tablets which are produced by most pharmaceutical manufacturers, including the State Pharmaceutical Manufacturing Corporation (SPMC) of Sri Lanka, contain a mixture of polymorphs A and C. However, there is some evidence to show that mebendazole polymorph C is the only form effective against the soil-transmitted helminths. This protocol describes a stratified, randomized, placebo-controlled trial that examined the efficacy of different mebendazole polymorphs produced by the SPMC in the treatment of hookworm infections.

DETAILED DESCRIPTION:
Mebendazole has three polymorphic forms, identified as A, B and C. All of them are in accord with the US Pharmacopeia specifications (USP XXI) but they have distinct physiochemical characteristics (Himmelreich et al, 1977) and different therapeutic activities in experimentally infected mice with Trichinella spiralis infections (Rodriguez-Caabeiro et al, 1987). The original mebendazole tablets which were used to treat human infections had more than 90% of polymorph C (Van den Bossche et al, 1982), but most pharmacopeias currently do not specify the proportion of polymorph C that a tablet of mebendazole should contain, and the assay specified for measurement of the active ingredient measures all polymorphs together. There is some evidence to show that unlike polymorph C, polymorph A is ineffective in the treatment of hookworm and whipworm infections (Charoenlarp et al, 1993). The State Pharmaceutical Manufacturing Corporation of Sri Lanka produces both 500 mg and 100 mg tablets of mebendazole according to specifications laid down in the US Pharmacopeia. These tablets contain a mixture of polymorphs A and C. It is possible that increasing the content of mebendazole polymorph C in single dose tablets may improve cure rates and egg reduction rates, especially against hookworm and whipworm infections, where much variation in efficacy has been observed.

ELIGIBILITY:
Inclusion Criteria:

* Necator americanus infection, as determined by examination of a single faecal smear, alone or with Ascaris lumbricoides or Trichuris trichiura

Exclusion Criteria:

* Children below the age of 2 years
* Pregnant women
* Individuals with diarrhea on day of treatment

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilanthi R de Silva, MD, Principal Investigator — Faculty of Medicine, University of Kelaniya, Sri Lanka
Locations (2):
- Sri Lanka (2):
  - Agalawatta Plantations PLC, Nivithigala, Sabragamuwa
  - Lellopitiya Estate, Hapugastenne Plantations PLC, Ratnapura, Sabragamuwa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In order to identify those with hookworm infections, all individuals living in 219 households, in 8 estate divisions in Ratnapura District known to have a high prevalence of hookworm, were recruited to the study after obtaining their written, informed consent. Each person was requested to provide one faecal sample.
Pre-assignment Details: Infants below the age of 2 years, pregnant women, and those with diarrhoea on the day of recruitment were excluded from the study.
Groups:
- Placebo: 70 were allocated to this arm and 49 were followed up in the post treatment.
- Mebendazole Polymorph A and C 500 mg: 70 were allocated and 53 were followed up in the post treatment.
- Mebendazole Polymorph C 500 mg: 74 were allocated and 48 were followed up in the post treatment.
Period: Overall Study
Arm/Group | Placebo | Mebendazole Polymorph A and C 500 mg | Mebendazole Polymorph C 500 mg
Started | 70 | 70 | 74
Completed | 49 | 53 | 48
Not Completed | 21 | 17 | 26
Not completed — Lost to Follow-up | 21 | 17 | 26

BASELINE CHARACTERISTICS:
Population: All those found positive for hookworm infection, from among the population screened at baseline
Groups:
- Placebo: Hookworm positive participants randomized to placebo
- Mebendazole Polymorph A and C 500 mg: Hookworm positive participants randomized to a single dose of Mebendazole polymorph A and C 500 mg
- Mebendazole Polymorph C 500 mg: Hookworm positive participants randomized to a single dose of Mebendazole polymorph C 500 mg
- Total: Total of all reporting groups
Arm/Group | Placebo | Mebendazole Polymorph A and C 500 mg | Mebendazole Polymorph C 500 mg | Total
Number analyzed (Participants) | 70 | 70 | 74 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 18 | 23 | 58
  Between 18 and 65 years | 49 | 48 | 47 | 144
  >=65 years | 4 | 4 | 4 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (18) | 36 (19) | 32 (18) | 34 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 40 | 114
  Male | 33 | 33 | 34 | 100
Region of Enrollment [Number; unit: participants]
  Sri Lanka | 70 | 70 | 74 | 214

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate
Description: Cure rate={(Number positive pretreatment - Number positive posttreatment)÷(Number positive pretreatment)}×100
Time Frame: Two weeks
Population: All participants who were hookworm positive at baseline, and who provided a faecal sample for examination at follow up.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Hookworm infected individual randomized to placebo
- Mebendazole Polymorph A and C 500 mg: Hookworm infected individuals randomized to a single dose of Mebendazole polymorph A and C 500 mg
- Mebendazole Polymorph C 500 mg: Hookworm infected individuals randomized to a single dose of Mebendazole polymorph C 500 mg
Arm/Group | Placebo | Mebendazole Polymorph A and C 500 mg | Mebendazole Polymorph C 500 mg
Number analyzed (Participants) | 49 | 53 | 48
percentage of participants | 16.3 | 28.3 | 18.8

2. Secondary Outcome: Faecal Egg Count Reduction 1 (FECR1)
Description: FECR1= {[(Arithmetic mean of pretreatment egg counts)-(arithmetic mean of posttreatment egg counts)]÷(arithmetic mean of pretreatment egg counts)}×100
Time Frame: Two weeks
Population: All participants who were hookworm positive at baseline, and who provided a faecal sample for examination at follow-up, were included in the analysis
Measure: Number; unit: percentage of eggs excreted
Groups:
- Mebendazole Polymorph C 500 mg: Hookworm positive participants randomized to a single dose Mebendazole polymorph C 500 mg
Arm/Group | Placebo | Mebendazole Polymorph A and C 500 mg | Mebendazole Polymorph C 500 mg
Number analyzed (Participants) | 49 | 53 | 48
percentage of eggs excreted | -6.6 | 86.1 | 84.5

3. Secondary Outcome: Faecal Egg Count Reduction 2 (FECR2)
Description: FECR2=〈Arithmetic mean {[(pretreatment egg count)-(posttreatment egg count)]÷(pretreatment egg count)}〉×100
Time Frame: Two weeks
Population: All participants who were hookworm positive at baseline, and who provided a faecal sample for examination at follow up were included in the analysis
Measure: Mean (Standard Deviation); unit: percentage of eggs excreted
Arm/Group | Placebo | Mebendazole Polymorph A and C 500 mg | Mebendazole Polymorph C 500 mg
Number analyzed (Participants) | 49 | 53 | 48
percentage of eggs excreted | -108.1 (557.5) | 66.2 (42.5) | 49.8 (82.6)

ADVERSE EVENTS:
Arm/Group | Placebo | Mebendazole Polymorph A and C 500 mg | Mebendazole Polymorph C 500 mg
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 0/74
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 0/74

LIMITATIONS AND CAVEATS:
Small sample size owing to limitation in available funds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Release after two years after completing trial